CLINICAL TRIAL: NCT01206959
Title: Clinical Test for Armed-used Blood Pressure Monitor With Preformed Cuff(Monitor When Being Inflated)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Liu Yi, Andon Health Co., LTD
Other Study IDs: AndonHealth 4
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Blood Pressure
Keywords: BP

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- monitor method: blood pressure monitor Cuff circumference:22cm-48cm
  stethoscopy Cuff circumference: 22cm-48cm

SUMMARY:
The purpose of this study is to monitor the blood pressure level of the patient using a blood pressure monitor which test the blood pressure level in inflating state . The cuff range in the study is 22cm-48cm

ELIGIBILITY:
Inclusion Criteria:

* cuff circumference:22cm-48cm

Exclusion Criteria:

* None

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hospital population, including patient and accompanies.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)